CLINICAL TRIAL: NCT04832386
Title: COMPLIANCE TO COMPRESSION GARMENTS AND RELATED FACTORS AMONG PATIENTS With BREAST CANCER-RELATED LYMPHEDEMA
Brief Title: COMPRESSION GARMENTS in BREAST CANCER-RELATED LYMPHEDEMA
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Banu Dilek, Principal investigator, Dokuz Eylul University
Other Study IDs: DokuzEU.Com.Garments
Record Dates: First submitted 2021-03-22; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most common cancer in women. It is an important health problem that has been increasingly encountered in recent years. With the advances in treatment, the survival time after breast cancer is prolonged, and as a result, many women face certain diseases during this period. One of these diseases, breast cancer-related lymphedema, is characterized by abnormal accumulation of protein-rich fluid in the interstitial tissue, which can occur at any time after breast cancer surgery or radiotherapy and is a major cause of morbidity. The aims of the treatment of lymphedema are to reduce edema, prevent the increase of edema, prevent infections, protect skin integrity, range of motion and limb functions. Complete Decongestive Therapy (CDT) is recommended by the International Society of Lymphology (ISL) as the international contemporary standard treatment for BCRL(breast cancer related lymphedema) treatment. CDT is a treatment method that includes manual lymph drainage (MLD), multilayer bandaging (Multilayer, short-stretch compression bandaging), exercise, skin care and compression garment. Compression garments, which are the most important component of the second phase of CDT, reduce the interstitial pressure of the extremity with the pressure they apply, and reduce capillary filtration and lymph production. Regular use of compression garments is very important during the treatment process. It is recommended that compression garments be worn during all waking hours. The success of compression garments is closely related to the patient's compliance with the treatment. Patients with lymphedema may need to wear compression garments for life. Wearing compression garments may have some difficulties for patients and this may affect compliance and adherence to treatment. The aim of this study is to investigate the compliance to compression garments and related factors among patients with breast cancer-related lymphedema.

DETAILED DESCRIPTION:
This study was planned as a cross-sectional study. Patients diagnosed with unilateral breast cancer-related lymphedema and recommended compression garments will be included in the study on a voluntary basis, after obtaining their written consent. Patients who have received a standard treatment and an education about the use of compression garments from a single center will be asked to answer our 28-question questionnaire about the use of compression garments. The patients will be asked whether compression garments were recommended or not, how long they have used compression garments, the type and model of the recommended compression garment, whether they can buy the recommended compression garment, how often it is changed, how long it is recommended to wear it during the day, whether it is used for the recommended time, how long wore during the day, the reasons for using and not using the garment. Compliance to compression garments and the factors affecting this will be questioned. Patients who use their garments for the recommended time and manner and those who do not will be compared in terms of these factors. Patients who used their garments for the recommended time and manner will be considered as compliant.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Diagnosed with breast cancer related lymphedema
* Having been prescribed compression garments

Exclusion Criteria:

* cognitive and / or psychiatric illness
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with breast cancer releated lymphedema
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
28-questionnaire about the use of compression garments | baseline
  Patients will be asked to answer our 28-questionnaire about the use of compression garments. Patients who used their garments for the recommended time and manner will be considered as compliant.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Dilek, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Erdinc Gunduz N, Sahin E, Dilek B, Ellidokuz H, Akalin E. Adherence to Compression Garment Wear and Associated Factors Among Patients with Breast Cancer-Related Lymphedema: A Pilot Study from a Turkish Tertiary Center. Lymphat Res Biol. 2022 Dec;20(6):665-670. doi: 10.1089/lrb.2021.0091. Epub 2022 Mar 3. PMID 35245100